CLINICAL TRIAL: NCT07195903
Title: Evaluation of Supracardiac Venous Angioplasty and Stenting on Ortho- Static Intolerance and Orthostatic Hypotension - The STANDUP Study
Brief Title: The STAND-UP Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-01; 25-01 (Other: St. Francis Hospital IRB)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Orthostatic Hypotension, Dysautonomic; Orthostatic Intolerance
MeSH Terms: conditions — Shy-Drager Syndrome; Orthostatic Intolerance | interventions — Angioplasty; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention (Experimental): Venous Angioplasty or stenting
  Interventions: Device: Angioplasty or stenting

INTERVENTIONS:
Device: Angioplasty or stenting — Jugular Vein Stenting
  Other Names: Venous Stenting

SUMMARY:
Orthostatic hypotension (OH) and orthostatic intolerance (OI) are common conditions where blood pressure drops when standing up, causing dizziness, fainting, or fatigue. These affect up to 30% of adults over 65 and raise risks for heart disease, stroke, kidney problems, and more. Current medications often don't fully help and can cause side effects like high blood pressure when lying down.

The STANDUP study tests a new approach: using a minimally invasive procedure to open narrowed veins above the heart (supracardiac veins) that may block blood flow back to the heart. We believe fixing these blockages could improve blood pressure control and reduce symptoms. This is a 2-year study enrolling 100 adults (age 18+) with OH or OI that hasn't improved with standard treatments or is worsened by lying-down high blood pressure.

What happens in the study? Participants get imaging (like X-rays and ultrasound) to check for vein narrowing. If needed, doctors use a thin tube (catheter) through a small skin puncture to inflate a tiny balloon (angioplasty) or place a small mesh tube (stent) to widen the veins. The procedure takes a few hours under local anesthesia, with monitoring for safety. Follow-up visits check symptoms, blood pressure, and quality of life at 2-4 weeks, 3 months, 6 months, 1 year, and 2 years.

Who can join?

Adults 18+ with diagnosed OH/OI not helped by meds. Must give informed consent. Not eligible if: Pregnant, breastfeeding, actively infected, or unable to take blood thinners.

Possible benefits: Better standing tolerance, fewer symptoms, improved daily life, less need for meds, and new knowledge on vein issues in OH/OI.

Risks: Rare but include bleeding, infection, stroke, vein clots, stent issues, radiation from imaging, or temporary symptom worsening. We'll monitor closely and report any problems.

This single-arm trial (no placebo group) will compare before-and-after results to see if the procedure helps. No study drug costs; covered by insurance or clinic. Led by Dr. Karthikeyan Arcot at St. Francis Hospital, Roslyn, NY. Contact for details.

ELIGIBILITY:
Inclusion criteria :

1. Age 18 years
2. Diagnosed orthostatic intolerance or orthostatic hypotension not responding to standard medical management or complicated by supine hypertension
3. Able to provide informed consent • Exclusion criteria:

1. Pregnancy or breastfeeding 2. Active infection 3. Coagulopathy or contraindication to anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | From enrollment to 6 months after
  Orthostatic blood pressures are measured and medication use is addressed

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan M Arcot, MD, Principal Investigator — St. Francis Hospital The Heart Center
Locations (1):
- St. Francis Hospital The Heart Center, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
Plan Description: Individual participant data (IPD) will not be shared with other researchers due to privacy concerns and the need to protect patient confidentiality, as well as the absence of specific funding or infrastructure to support data sharing at this time.